CLINICAL TRIAL: NCT05657548
Title: Study of Sagittal Pelvic Statics in the Sitting Position in Children With Cerebral Palsy
Acronym: SPS-PC
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2022/CL-01; ANSM (Other: 2022-A01466-37)
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy Infantile
Keywords: Spine; Child; Adolescent; Pelvis; Postural Balance; Posture; Radiography
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Child with Cerebral Palsy: Children and adolescents from 4 to 17 years old with cerebral palsy GMFCS III, IV or V followed in the Physical Medicine and Rehabilitation Department, Children's Rehabilitation Unit of the University Hospital of Nîmes (Carémeau Hospital)
  Interventions: Radiation: spine and pelvis radiography

INTERVENTIONS:
Radiation: spine and pelvis radiography — X-ray of the spine and pelvis from the front and the side will be performed under the standardized conditions that we put in place: in a sitting position on a specific modular chair.

SUMMARY:
Cerebral palsy is the leading cause of motor disability in children. Children with little or no walking (GMFCS III, IV and V) represent 43% of children with cerebral palsy, the majority of whom present pelvic and spinal deformities in the frontal and sagittal planes. However, sagittal pelvic spinal statics have been little studied, especially in the sitting position, which is the functional position of these children.

Moreover, there are currently no recommendations on how to perform follow-up radiographs of the spine in children who do not walk much.

A better understanding of pelvic and sagittal spinal statics would help prevent deformities and their complications.

Standardizing the method of performing pelvic-spinal radiographs in the sitting position will make monitoring of spinal statics more reliable.

ELIGIBILITY:
Inclusion Criteria:

* Child or adolescent aged 4 to 17 years
* Child or adolescent with cerebral palsy GMFCS III, IV or V
* Child or adolescent whose parents, or the child if possible, have given free, informed and written consent
* Child or adolescent affiliated or beneficiary of a health insurance plan

Exclusion Criteria:

* Child or adolescent with history of spinal surgery
* Child or adolescent with parents unable to give consent
* Child or adolescent participating in a therapeutic research study (RIPH 1 or drug study)
* Child or adolescent in an exclusion period determined by another study
* Child or adolescent under court protection, guardianship or curatorship
* Pregnant, parturient or breastfeeding patient

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents from 4 to 17 years old with cerebral palsy GMFCS III, IV or V followed in the Physical Medicine and Rehabilitation Department, Children Rehabilitation Unit of the CHU of Nîmes
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Evolution of the sagittal spinal statics in the sitting position | At baseline
  measurement of pelvic incidence (normal values between 35 and 85 degrees)
Evolution of the sagittal spinal statics in the sitting position | At baseline
  sacral slope (angle of inclination of the sacral plateau in profile to the horizontal (degrees))
Evolution of the sagittal spinal statics in the sitting position | At baseline
  pelvic version (angle between the vertical and the line joining the center of the femoral heads with the middle of the sacral plateau (in degrees))
Evolution of the sagittal spinal statics in the sitting position | At baseline
  lordoses cervicales (in degrees)
Evolution of the sagittal spinal statics in the sitting position | At baseline
  lumbar lordosis (in degrees)
Evolution of the sagittal spinal statics in the sitting position | At baseline
  thoracic kyphosis (in degrees)
Evolution of the sagittal spinal statics in the sitting position | At baseline
  Cobb angle (if scoliosis) (curvature greater than 10 degrees : definition of scoliosis; between 10 and 15 degree: benign scoliosis; between 15 and 35 degrees: moderate scoliosis; curvature greater than 35 degrees: significant scoliosis.)

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No